CLINICAL TRIAL: NCT03246308
Title: Investigation of Vitamin Levels During Phototherapy
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Benedikt Weber, MD PhD, Medical University of Vienna
Other Study IDs: 1462/2017
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-05

CONDITIONS: Phototherapy Complication
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Phototherapy — Taking blood sample.

SUMMARY:
Research project in which blood samples of patients undergoing UVB phototherapy for the treatment of different cutaneous diseases will be investigated for changes of folate levels and further vitamins over the course of treatment.

DETAILED DESCRIPTION:
UVB phototherapy is used to treat a plethora of different dermatoses with a favorable side effect profile compared to systemic alternatives. One rarely mentioned issue related to phototherapy is the question of whether it holds potential to decrease folate serum levels, which is of particular interest to women of childbearing age, as birth defects, such as neural tube defects (NTD), cardiac defects, and facial clefting have all been noted to be increased in women with folate deficiency. Several studies, involving different patient groups and modes of phototherapy, have investigated the changes of folate levels throughout therapy showing mixed results. While two small open studies from Egypt showed a significant reduction of folate levels after 24 and 18 / 36 exposures (1-2), several other studies failed to show a significant change (3-6). In addition, there are also conflicting data on the influence of UVB phototherapy on vitamin D, vitamin B12 and homocysteine levels. Therefore, the presented prospective trial aims at investigating the changes of these vitamins during a routine course of phototherapy. The study will focus on the following specific aims: Measure the levels of folate as well as the levels of further vitamin parameters (including homocysteine, 25-OH-vitamin D3, 1,25-OH-vitamin D3, holotranscobalamin and methylmalonic acid) before and during phototherapy (at baseline, after 12, 24 and 36 exposures and/or at the end of treatment)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing UVB phototherapy (narrowband UVB or broadband UVB)
* Male and female participants minimum 18 years old
* Written informed consent by the participant after information about the research project

Exclusion Criteria:

* Regular sunbed use
* Underlying disease with abnormal folate metabolism (e.g. thalassemia)
* Age below 18 years
* Patients who will not be able to attend regularly for treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing UVB therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Folate level | 3 years
  The change of the folate levels will be measured at baseline and at the end of phototherapy.
vitamin D level | 3 years
  The change of vitamin D levels will be measured at baseline and at the end of phototherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No